CLINICAL TRIAL: NCT05480150
Title: Chinese Longitudinal and Systematic Study of Bioplar Disorder
Acronym: CLASS-BD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Principal Investigator, Hu ShaoHua, Head of Department of Psychaitry , First Affiliated Hospital of Zhejiang University, First Affiliated Hospital of Zhejiang University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT20210291B-R1
Record Dates: First submitted 2022-07-28; First posted 2022-07-29 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: Major Depressive Disorder; Bipolar Disorder, Mixed; Affective; Disorder, Organic
Keywords: Major Depressive Disorder; Bipolar Disorder; Affective Disorder; Gut-Brain Axis
MeSH Terms: conditions — Depressive Disorder, Major; Bipolar Disorder; Mood Disorders | interventions — Escitalopram; Quetiapine Fumarate; Lurasidone Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- bipolar disorder (Experimental): Patients with BD depressive episode received standard treatment with quetiapine fumarate tablets, starting from 50mg/ night, titrated to a therapeutic dose of 300-400mg/ night within 10 days, and maintained treatment for 4 weeks. According to the patient's condition, patients with BD depressive episode could receive another standard treatment with lurasidone, starting from 20mg/ night, titrated to a therapeutic dose of 40mg/ night within 6 days, and maintained treatment for 4 weeks. Adverse reactions and changes in condition of all patients were recorded
  Interventions: Drug: Quetiapine Fumarate Tablets; Drug: Lurasidone
- major depressive disorder (Experimental): MDD depressive episode patients received standard treatment with escitalopram oxalate tablets, starting from 5mg/ day once, titrated to a therapeutic dose of 10-20mg/ day within 1 week, and maintained treatment for 4 weeks
  Interventions: Drug: Escitalopram Oxalate Tablets
- healthy control (No Intervention): no interventions

INTERVENTIONS:
Drug: Escitalopram Oxalate Tablets — Starting at 5mg qn, the treatment dose was titrated to 10-20mg qn within 1 week and maintained for 4 weeks
  Other Names: Lexapro
  Arms: major depressive disorder
Drug: Quetiapine Fumarate Tablets — Starting at 50mg qn, the treatment dose was titrated to 300-400mg qn within 10 days, and maintained the treatment for 4 weeks.
  Other Names: Seroquel
  Arms: bipolar disorder
Drug: Lurasidone — Starting at 20mg qn, the treatment dose was titrated to 40mg qn within 6 days,and maintained the treatment for 4 weeks.
  Other Names: Latuda
  Arms: bipolar disorder

SUMMARY:
Affective disorders (mainly including major depressive disorder and bipolar disorder) are common, chronic and highly disabling mental disorders, which lack of objective biological markers. It is believed that genetic and environmental factors are involved in the development of affective disorders. Gut microbes can affect the function of brain neural circuits by mediating metabolic, immune, endocrine and autonomic changes along the brain-gut axis. The brain can also regulate intestinal microbes through endocrine, neural structure, neurogenic exosomes and other pathways. Based on the brain-gut axis, this study intends to establish a large cohort of affective disorders, and screen out efficient and convenient biomarkers for clinical diagnosis and efficacy prediction by studying key indicators such as intestinal microbes, serum metabolites and immune indexes, brain-derived exosomes, and brain functional imaging.

DETAILED DESCRIPTION:
Mental health is a major public health problem affecting the whole social and economic development. According to a 2019 report in The Lancet Psychiatry, the weighted lifetime prevalence of mental disorders (excluding dementia) in China is 16.6%, with the lifetime prevalence of emotional disorders as high as 7.4%.Affective disorders (mainly including depression and bipolar disorder) are common, chronic and highly disabling mental disorders.Back in 2008, the World Health Organization listed MDD（Major Depressive Disorder） as one of the three major contributors to the overall global burden of disease. It is expected that by 2030, the number of MDD patients will exceed the total number of cardiovascular disease patients combined and become the leading cause of disability in the world.

At present, the diagnostic criteria of mental disorders, including DSM-5 and ICD-11, still mainly rely on the evaluation of symptoms, lacking objective and intuitive biomarkers. Therefore psychiatrists are prone to disagreement in diagnosis and treatment of diseases, which is a realistic bottleneck hindering the development of psychiatry. The differential diagnosis of MDD and BD depressive episodes is an unavoidable clinical challenge, which often leads to misdiagnosis and affects the treatment and prognosis of the disease. Therefore, it is one of the important directions for the development of brain science to strengthen scientific research in the field of mental health, especially to explore the mechanism of disease occurrence and development, develop objective new auxiliary diagnostic technologies and innovate precise treatment strategies around major emotional disorders. It is believed that genetic and environmental factors are involved in the development of affective disorders. Gut microbes can affect the function of brain neural circuits by mediating metabolic, immune, endocrine and autonomic changes along the brain-gut axis. The brain can also regulate intestinal microbes through endocrine, neural structure, neurogenic exosomes and other pathways. This study based on brain - im axis, intends to create an emotional disorder large queue, through the study of gut microbes (diversity and abundance of species), serum metabolites, and immune index, brain outside source sex secretion, brain imaging and other key indicators, select high efficiency and convenient for clinical diagnosis and curative effect of prediction of biomarkers.

ELIGIBILITY:
Inclusion Criteria:

1. Both biological parents are Han nationality;
2. Aged 16-65;
3. The subjects met the clinical diagnostic criteria of DSM-5 for depressive episodes of MDD/BD;
4. Did not take any immunomodulatory preparations within 1 month before enrollment;
5. No clear history of respiratory tract, urinary system, digestive system infection within 1 month before enrollment;

Exclusion Criteria:

1. Those with schizophrenia spectrum, neurodevelopmental disorder, dementia, memory impairment or other cognitive impairment that meet the DIAGNOSTIC criteria of DSM-5;
2. Mental disorders caused by substance abuse (alcohol, drugs, etc.), patients suffering from serious physical diseases and immune system diseases, such as diabetes, thyroid diseases, hypertension, heart disease, liver and kidney dysfunction, autoimmune diseases, etc.;
3. Had received medication (such as antidepressants, antipsychotics, mood stabilizers, etc.) within 1 month before enrollment;
4. those who had used ECT before enrollment;
5. Currently have serious suicidal thoughts or behaviors, or serious excitement;
6. those who cannot follow the doctor's advice or have no guardian;
7. pregnant or breast-feeding women, or those who plan to become pregnant;
8. Contraindications to MRI examination;
9. Other conditions that the researcher considers inappropriate for inclusion.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10000 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale(MADRS) | 0 ~16 weeks
  MADRS score is to evaluate the degree of depression, and the higher score means severer depression.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
Arms and interventions can be shared, while the clinical data will not be shared

REFERENCES:
- [Derived] Tang A, Chen Y, Ding J, Li Z, Xu C, Hu S, Lai J. Gut microbiota remodeling and sensory-emotional functional disruption in adolescents with bipolar depression. J Transl Med. 2025 Oct 14;23(1):1083. doi: 10.1186/s12967-025-07152-4. PMID 41088296